CLINICAL TRIAL: NCT05183321
Title: Treatment of Periodontal Disease in Patients With Alzheimer's Disease: Randomized Controlled Trial
Brief Title: Treatment of Periodontal Disease in Patients With Alzheimer's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KQCLLAD001
Record Dates: First submitted 2021-12-26; First posted 2022-01-10 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-04

CONDITIONS: Periodontitis; Alzheimer Disease; Dementia
MeSH Terms: conditions — Periodontitis; Alzheimer Disease; Dementia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control Group (No Intervention): Group will not receive treatment: periodontal therapy
- Periodontal therapy (Experimental): Group will receive treatment: periodontal therapy
  Interventions: Procedure: periodontal therapy

INTERVENTIONS:
Procedure: periodontal therapy — periodontal cleaning
  Arms: Periodontal therapy

SUMMARY:
The main objective of this study is to evaluate the effect of periodontal therapy in in subjects with a clinical diagnosis of mild to moderate AD dementia.

DETAILED DESCRIPTION:
This is a randomized, controlled study that will assess the effects of periodontal therapy in subjects with probable AD dementia according to the National Institute on Aging-Alzheimer's Association (NIA-AA) criteria. The study will enroll approximately 190 generally healthy male and female subjects ≥55 and ≤80 years of age. Enrolled subjects must have a documented diagnosis of mild to moderate AD dementia. The subject should not have other conditions or brain imaging abnormalities that can explain the symptoms of dementia. All subjects will be encouraged to have LPs (during screening, week 28 and week 52) in the absence of medical conditions that can increase the risk of the procedure in the opinion of the Investigator. Cerebrospinal fluid (CSF) and blood will be analyzed for measurements of biomarkers of AD and neuroinflammation, PiB-PET will be done for assessment of AD. A subset of sites will monitor subjects for clinical evidence of periodontitis at baseline, 28 and 52 weeks.

The study will consist of 3 phases: a screening phase of up to 8 weeks, a treatment phase of up to 52 weeks, and a safety follow-up phase of 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subject has primary school education or above.
* Subject has probable AD dementia according to the NIA-AA criteria.
* Subject has brain MRI scan consistent with the diagnosis of AD performed during the screening period. Computed Tomography scan can be used only if the subject has an absolute contraindication for MRI.
* Subject has a Modified Hachinski score ≤4 at screening.
* Subject has an MMSE score ≥15 at screening.
* Subjects with background symptomatic therapy with acetylcholine esterase inhibitors, and/or memantine, are allowed as long as the dose has been stable for 90 days prior to screening and no changes are planned during the study.
* Subject has a primary caregiver willing to accept responsibility for supervising the treatment (e.g., administering study drug) and assessing the condition of the subject throughout the study in accordance with all protocol requirements.
* Subject has body mass index <38 kg/m2 at Screening

Exclusion Criteria:

* Subject has imaging consistent with a dementia diagnosis other than AD.
* Subject has had an increase or restoration of cognition based on medical history.
* Subject with history or current evidence of major psychiatric illness such as schizophrenia, bipolar disorder, or major depressive disorder that may interfere with the patient's ability to perform the study and all assessments. NOTE: Mild depression or depressive mood arising in the context of AD are not criteria for exclusion. The use of anti-depressants or the use of anti epileptic medication for non seizure-related treatment is allowed if the dose has remained stable for at least 60 days prior to enrollment.
* Subject is fitted with pacemakers (except for new compatible products), large ferromagnetic implants, or implanted electronic devices such as cochlear implants, magnetic metal drug infusion pumps, nerve stimulators, diaphragmatic stimulators and injection pumps, physiological stimulators, and cardiac mechanical valves.
* Subject has magnetic metal foreign body or prosthesis in eye, magnetic metal joint or ferromagnetic foreign body in body.
* Subject has epilepsy or claustrophobia.
* Subject had received antibiotics or periodontal treatment within the last 6 months.
* Subject had taken aspirin, warfarin and other anticoagulant drugs in the last 6 months.
* Subject has any of the following laboratory findings at screening:

  1. Coagulation disorders.
  2. Hemoglobin ≤10 g/dl.
  3. Poorly controlled diabetes as defined by hemoglobin A1C (HbA1C) >8.
  4. Positive blood screen for Human Immunodeficiency Virus (HIV 1 and 2), Hepatitis B surface antigen (HBsAg), or Hepatitis C virus antibodies (HCV-Ab) at Screening.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale-Cognitive Subscale 11 (ADAS-Cog 11) | 52 weeks
  Mean change in Alzheimer's Disease Assessment Scale-Cognitive Subscale 11 (ADAS-Cog 11) from baseline to the end of treatment period. ADAS-Cog 11 measures cognitive functions and non-cognitive functions such as mood and behavior. Total scores range from 0-70, with higher scores (≥ 18) indicating greater cognitive impairment. ADAS-Cog 11 score increases by 2-4 points per year on average in subjects with mild to moderate Alzheimer's Disease. A treatment period of 52 weeks was selected to allow sufficient time to demonstrate at least 2.5 points difference between active treatment and placebo on ADAS-Cog 11 at the end of the treatment period.
ADCS-ADL | 52 weeks
  Change in Alzheimer's Disease Cooperative Study Group-Activities of Daily Living (ADCS-ADL)

SECONDARY OUTCOMES:
MMSE | 52 weeks
  Change in Alzheimer's Disease Cooperative Study Group-Activities of Daily Living Change in Mini-Mental State Examination (MMSE).
MoCA | 52 weeks
  Change in Montreal Cognitive Assessment Scale

OTHER OUTCOMES:
PiB-PET | 52 weeks
  Change in PiB-PET
Tau-PET | 52 weeks
  Change in Tau-PET
Tau levels in cerebrospinal fluid | 52 weeks
  Change in Tau levels in cerebrospinal fluid
Aβ levels in cerebrospinal fluid | 52 weeks
  Change in Aβ levels in cerebrospinal fluid
Magnetic resonance imaging | 52 weeks
  Change in magnetic resonance imaging
Periodontal (or gum) pocket depth | 52 weeks
  Change in periodontal (or gum) pocket depth

CONTACTS AND LOCATIONS:
Overall Officials: Lili Chen, Study Chair — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology